CLINICAL TRIAL: NCT04881032
Title: Phase I/II Study of AGuIX Nanoparticles With Radiotherapy Plus Concomitant Temozolomide in the Treatment of Newly Diagnosed Glioblastoma
Brief Title: AGuIX Nanoparticles With Radiotherapy Plus Concomitant Temozolomide in the Treatment of Newly Diagnosed Glioblastoma
Acronym: NANO-GBM
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Collaborators: Ministry for Health and Solidarity, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-004552-15
Record Dates: First submitted 2021-04-30; First posted 2021-05-11 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — AGuIX; Radiotherapy; Temozolomide

STUDY DESIGN:
Intervention Model Description: Phase 1 : dose escalation Phase 2 : randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AGuIX + chemoradiotherapy (radiotherapy + temozolomide) (Experimental): addition of AGuIX nanoparticles to standard radiotherapy and concomitant treatment by temozolomide (TMZ) for patients of phase I and patients randomized in experimental arm of phase II
  Interventions: Drug: Polysiloxane Gd-Chelates based nanoparticles (AGuIX); Radiation: radiotherapy; Drug: Temozolomide
- chemoradiotherapy (radiotherapy + temozolomide) (Sham Comparator): standard of care : chemoradiotherapy (radiotherapy + temozolomide) for patients randomized in control arm of phase II
  Interventions: Radiation: radiotherapy; Drug: Temozolomide

INTERVENTIONS:
Drug: Polysiloxane Gd-Chelates based nanoparticles (AGuIX) — Four intravenous injections of AGuIX will be delivered. Phase I : Three dose levels may be explored 50 mg/kg, 75 mg/kg and 100 mg/ kg. Phase II : recommended dose
  Arms: AGuIX + chemoradiotherapy (radiotherapy + temozolomide)
Radiation: radiotherapy — 60 Gy in 6 weeks
Drug: Temozolomide — Concomitant chemotherapy consists of temozolomide (TMZ) at a dose of 75 mg per square meter per day, given 7 days per week from the first day of radiotherapy until the last day of radiotherapy.
  After a 4 week break after concomitant treatment, patient were then received up to 6 cycles of adjuvant TMZ according to the standard 5-day schedule every 28 days .

SUMMARY:
This is a phase I/II clinical trial evaluating the association of AGuIX nanoparticles with radiotherapy plus concomitant Temozolomide in the treatment of newly diagnosed glioblastoma.

The primary objectives of this study were to determine the recommended dose of AGuIX in combination with radiotherapy and TMZ during the concomitant radiochemotherapy period (phase I) and to estimate the efficacy of the combination radiochemotherapy + AGuIX (recommended dose), measured by the 6-month progression-free survival rate (PFS) (phase II)

Three dose levels of intravenous AGuIX nanoparticles will be explored: 50 mg/kg, 75 mg/kg and 100 mg/kg.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of grade IV glioblastoma (biopsy or partial surgery)
* Patient not operated or partial resection
* KPS superior to 70%
* Age between 18 years old and 75 years old
* Life expectancy superior to 6 months
* Platelets superior to 100,000 / mm3
* PNN superior to 1500 / mm3
* Hb superior to 10 g / dL
* Creatinine superior to 1.5 times the upper normal limit or clearance according to Cockcroft-Gault superior to 50 mL / min
* Liver function (GGT, PAL, ASAT, ALAT, bilirubin) superior to 1.5 times the upper normal limit
* For patients receiving treatment with corticosteroids, treatment with corticosteroids must be at a stable or decreasing dose for at least 14 days before inclusion
* Patient able to swallow and retain oral medication
* Negative serum pregnancy test within 7 days before the first administration of treatment for women
* Women of childbearing potential and men whose partners are of childbearing potential must agree to use, themselves or their partners, an approved method of contraception throughout the treatment and at least 6 months after the last administration of study treatment.
* Obtaining signed informed consent from the patient
* Patient affiliated to a social security regimen

Exclusion Criteria:

* prior brain radiotherapy
* prior chemotherapy (including implants containing carmustine (Gliadel®) or immunotherapy (vaccination included)
* Any contraindication to TMZ listed in the SPCs
* History of major intestinal resection which may modify the absorption of oral drugs according to the judgment of the investigator
* Diagnosed inflammatory bowel disease (Crohn disease or ulcerative colitis)
* Diarrhea superior to grade 2 CTCAE (whatever the cause)
* Current or recent treatment with another investigational drug or participation in another therapeutic clinical trial (within 30 days of inclusion).
* History of other cancer in the 5 years preceding inclusion, except for basal cell carcinomas of the skin and in situ carcinomas of the cervix
* Pregnant or breastfeeding women
* Contraindication to MRI or gadolinium injection
* History of severe anaphylactic reactions due to the injection of gadolinium-based contrast product (dotarem, etc.)
* Patient under guardianship or curatorship
* History of nephropathy
* Psychological disorder or social or geographic reasons that may compromise medical monitoring of the trial or compliance with treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
The recommended dose (phase I) of AGuIX in combination with TMZ and and radiotherapy during the radio-chemotherapy period | during 6 weeks after the first injection of AGuIX
  Only toxicities occurring during concomitant radiochemotherapy will be considered for the evaluation of Dose Limiting Toxicity radiotherapy during the radio-chemotherapy period is defined as the highest dose tested in which the % of dose-limiting toxicities (DLT) is less than 33%. DLT is defined as any grade 3-4 toxicity according to the NCI CTCAE v5.0 classification, except alopecia, nausea, and vomiting which can be quickly controlled with appropriate measures.
6-month Progression Free Survival (PFS) rate (phase II) | 6 months from the start of treatment

SECONDARY OUTCOMES:
Pharmacokinetic Cmax of AGuIX | Day 0 , Day 7, Day 14
  maximal plasma concentration (Cmax) of AGuIX
Pharmacokinetic Tmax of AGuIX | Day 0 , Day 7, Day 14
  time of maximal plasma concentration (Tmax) of AGuIX
Pharmacokinetic AUC of AGuIX | Day 0 , Day 7, Day 14
  Area Under the Curve (AUC) of AGuIX
Pharmacokinetic t1/2 of AGuIX | Day 0 , Day 7, Day 14
  pharmacokinetic term half-life (t1/2) of AGuIX
distribution of AGuIX | after the first and last injection of AGuIX, Week 0 and Day 14
  measure of RMI contrast enhancement in tumor and healthy tissue
Overall Survival | from the start of treatment to death, up to 24 months
Progression Free Survival (PFS) | from the start of treatment to progression, up to 24 months
Toxicity (CTCAE criteria) | from baseline to 30 days after treatment (concomitant and adjuvant treatment) (week 35)
  according to NCI Common Toxicity Criteria for Adverse Effect (CTCAE) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Juliette Moreau, Md, Principal Investigator — Centre Jean Perrin
Locations (9):
- France (9):
  - CHU de Brest, Brest
  - Centre Jean Perrin, Clermont-Ferrand
  - CHU de Grenoble, Grenoble
  - Centre Léon Berard, Lyon
  - Hospices Civils de Lyon, Lyon
  - Hôpital La Pitié Salpetrière, Paris
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Institut de Cancérologie Strasbourg Europe, Strasbourg
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] Thivat E, Casile M, Moreau J, Molnar I, Dufort S, Seddik K, Le Duc G, De Beaumont O, Loeffler M, Durando X, Biau J. Phase I/II study testing the combination of AGuIX nanoparticles with radiochemotherapy and concomitant temozolomide in patients with newly diagnosed glioblastoma (NANO-GBM trial protocol). BMC Cancer. 2023 Apr 15;23(1):344. doi: 10.1186/s12885-023-10829-y. PMID 37060055